CLINICAL TRIAL: NCT03696459
Title: A Double-blind, Randomized, Placebo-controlled, 4-Period Cross-over Study to Evaluate the Effect of JNJ-53718678 on the Cardiac Repolarization Interval in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Effect of JNJ-53718678 on the Cardiac Repolarization Interval in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CR108519; 2018-000878-30 (EudraCT Number); 53718678RSV1009 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-10-03; First posted 2018-10-04 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Healthy
MeSH Terms: interventions — JNJ-53718678; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Part 1 (Dose Escalation): Panel 1 (Experimental): Participants will receive single oral dose of JNJ-53718678, 2000 milligram (mg) suspension or matching placebo on Day 1, under fasted conditions.
  Interventions: Drug: JNJ-53718678, 2000 mg; Drug: JNJ-53718678 Placebo
- Part 1 (Dose Escalation): Panel 2 (Experimental): Participants will receive single oral dose of JNJ-53718678, of maximum 3000 mg suspension or matching placebo on Day 1, under fasted conditions.
  Interventions: Drug: JNJ-53718678, 3000 mg; Drug: JNJ-53718678 Placebo
- Part 1 (Dose escalation): Panel 3 (Experimental): Participants will receive single oral dose of JNJ-53718678 4500 mg suspension (this dose may be used in Part 2, Treatment F) or matching placebo on Day 1, under fasted condition.
  Interventions: Drug: JNJ-53718678, 4500 mg or Dose to be decided; Drug: JNJ-53718678 Placebo
- Part 1 (Dose Escalation): Panel 4 (Optional) (Experimental): Participants will receive single oral dose of JNJ-53718678 (dose to be decided [this dose may be used in Part 2, Treatment F]) suspension or matching placebo on Day 1, under fasted condition, if 4500 mg dose in Panel 3 is considered safe and tolerable and if pharmacokinetic data require further dose escalation to reach the target exposure.
  Interventions: Drug: JNJ-53718678, 4500 mg or Dose to be decided; Drug: JNJ-53718678 Placebo
- Part 2 Group 1: Treatment Sequence EHFG (Experimental): Participants will receive single oral dose of JNJ-53718678, 500 mg suspension with single oral dose of moxifloxacin placebo and JNJ 53718678 placebo (Treatment E) in Period 1, then participants will receive single oral dose of moxifloxacin 400 mg with single oral dose of JNJ-53718678 placebo (Treatment H) in Period 2 then will receive single oral dose of JNJ-53718678, 4500 mg (dose will be based on review of safety, tolerability, and PK data obtained in Part 1 [either from Panel 3 or 4], this dose may be lower/higher) suspension with single oral dose of moxifloxacin placebo (Treatment F) in Period 3 followed by single oral dose of JNJ-53718678 placebo with single oral dose of moxifloxacin placebo (Treatment G) in Period 4, on Day 1 of each treatment period. There will be a washout period of at least 7 days between study drug intake in subsequent treatment periods.
  Interventions: Drug: JNJ-53718678, 4500 mg or Dose to be decided; Drug: JNJ-53718678 500 mg; Drug: JNJ-53718678 Placebo; Drug: Moxifloxacin 400 mg; Drug: Moxifloxacin Placebo
- Part 2 Group 2: Treatment Sequence FEGH (Experimental): Participants will receive Treatment F in Period 1, then Treatment E in Period 2, then Treatment G in Period 3 followed by Treatment H in Period 4 on Day 1 of each treatment period.
  Interventions: Drug: JNJ-53718678, 4500 mg or Dose to be decided; Drug: JNJ-53718678 500 mg; Drug: JNJ-53718678 Placebo; Drug: Moxifloxacin 400 mg; Drug: Moxifloxacin Placebo
- Part 2 Group 3: Treatment Sequence GFHE (Experimental): Participants will receive Treatment G in Period 1, then Treatment F in Period 2, then Treatment H in Period 3 followed by Treatment E in Period 4 on Day 1 of each treatment period.
  Interventions: Drug: JNJ-53718678, 4500 mg or Dose to be decided; Drug: JNJ-53718678 500 mg; Drug: JNJ-53718678 Placebo; Drug: Moxifloxacin 400 mg; Drug: Moxifloxacin Placebo
- Part 2 Group 4: Treatment Sequence HGEF (Experimental): Participants will receive Treatment H in Period 1, then Treatment G in Period 2, then Treatment E in Period 3 followed by Treatment F in Period 4 on Day 1 of each treatment period.
  Interventions: Drug: JNJ-53718678, 4500 mg or Dose to be decided; Drug: JNJ-53718678 500 mg; Drug: JNJ-53718678 Placebo; Drug: Moxifloxacin 400 mg; Drug: Moxifloxacin Placebo

INTERVENTIONS:
Drug: JNJ-53718678, 2000 mg — Participants will be administered JNJ-53718678, 2000 mg as oral suspension in Part 1 (Panel 1).
  Arms: Part 1 (Dose Escalation): Panel 1
Drug: JNJ-53718678, 3000 mg — Participants will be administered JNJ- 53718678, 3000 mg as oral suspension in Part 1 (Panel 2).
  Arms: Part 1 (Dose Escalation): Panel 2
Drug: JNJ-53718678, 4500 mg or Dose to be decided — Participants will be administered JNJ-53718678, 4500 mg as oral suspension in Part 1 (Panel 3). If this dose is considered safe and tolerable and if pharmacokinetic data require further dose escalation, then participants will receive JNJ-53718678 (Dose to be decided) in Part 1 (Panel 4). This dose (either from Panel 3 or Panel 4 ) will be used in Part 2 (Dose may be lower/higher based on review of safety, tolerability, and PK data obtained in Part 1).
  Arms: Part 1 (Dose Escalation): Panel 4 (Optional); Part 1 (Dose escalation): Panel 3; Part 2 Group 1: Treatment Sequence EHFG; Part 2 Group 2: Treatment Sequence FEGH; Part 2 Group 3: Treatment Sequence GFHE; Part 2 Group 4: Treatment Sequence HGEF
Drug: JNJ-53718678 500 mg — Participants will be administered JNJ-53718678, 500 mg as oral suspension in Part 2.
  Arms: Part 2 Group 1: Treatment Sequence EHFG; Part 2 Group 2: Treatment Sequence FEGH; Part 2 Group 3: Treatment Sequence GFHE; Part 2 Group 4: Treatment Sequence HGEF
Drug: JNJ-53718678 Placebo — Participants will be administered JNJ-53718678 matching placebo in Part 1 and 2.
Drug: Moxifloxacin 400 mg — Participants will be administered moxifloxacin 400 mg as capsule in Part 2.
  Arms: Part 2 Group 1: Treatment Sequence EHFG; Part 2 Group 2: Treatment Sequence FEGH; Part 2 Group 3: Treatment Sequence GFHE; Part 2 Group 4: Treatment Sequence HGEF
Drug: Moxifloxacin Placebo — Participants will be administered moxifloxacin matching placebo in Part 2.
  Arms: Part 2 Group 1: Treatment Sequence EHFG; Part 2 Group 2: Treatment Sequence FEGH; Part 2 Group 3: Treatment Sequence GFHE; Part 2 Group 4: Treatment Sequence HGEF

SUMMARY:
The purpose of this study is to assess the effect of JNJ-53718678 on QT interval corrected for heart rate (QTc) changes using exposure response analysis in healthy adult participants (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a Body mass index (BMI) between 18 and 30 kilogram per square meter (kg/m^2) (inclusive), and body weight not less than (<) 50 kg at screening
* Participants must have a blood pressure between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic at screening
* Participants must have a 12-lead electrocardiogram (ECG) consistent with normal cardiac conduction and function at screening, including: a) Normal sinus rhythm (heart rate (HR) between 45 and 100 beats per minute (bpm), inclusive); b) QT interval corrected for HR according to Fridericia's formula (QTcF) between 350 milliseconds (ms) and 430 ms for male participants, and between 350 ms and 450 ms for female participants (inclusive); c) QRS interval of ECG <110 ms; d) PR interval of the ECG less-than or equal to (<=) 200 ms; e) Morphology consistent with healthy cardiac conduction and function
* A female participant must be of non-childbearing potential, defined as: a) Postmenopausal or b) Permanently sterile
* A female participant must have a negative serum beta-human chorionic gonadotropin (b-hCG) pregnancy test at screening and a negative urine pregnancy test (except if postmenopausal) on Day -1 (or Day -2 in the first treatment period in Part 2)

Exclusion Criteria:

* Participants has a history of current clinically significant medical illness or certain laboratory abnormalities at screening
* Participant has a history of hepatitis A virus immunoglobulin M (IgM) antibody, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody positive, or other clinically active liver disease, or tests positive for hepatitis A virus IgM antibody, HBsAg or HCV antibody at screening
* Participants with unusual T wave morphology (such as bifid T wave) likely to interfere with QTc measurements
* Participants with a past history of heart arrhythmias or with a history of risk factors for Torsade de Pointes syndrome (for example, hypokalemia or family history of short/long QT syndrome, or sudden unexplained death at a young age [<=40 years], drowning or sudden infant death in a first degree relative [that is, sibling, offspring, or biological parent])
* Participants with any skin condition likely to interfere with ECG electrode placement or adhesion

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Part 2: Placebo-Corrected Change from Baseline in QT Interval Corrected for Heart Rate (QTc) for JNJ-53718678 | Baseline and Day 1
  Placebo-corrected change from baseline in QT interval corrected for heart rate (QTc) will be determined. The mean change from baseline in QTc in placebo treatment will be subtracted from the mean change from baseline in JNJ-53718678 treatment at the same time point to generate placebo-corrected change from baseline in QTc, which will be presented.

SECONDARY OUTCOMES:
Part 1: Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Approximately up to 9 weeks
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Part 2: Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Approximately up to 12 weeks
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Part 1: Change from Baseline in QTc Interval | Baseline, 3, 24, 72 hours and at follow-up (10-14 days postdose)
  The QT interval corrected for heart rate (QTc interval) using Fridericia method will be measured by electrocardiograms (ECG).
Part 1: Change from Baseline in Heart Rate (HR) | Baseline, 3, 24, 72 hours and at follow-up (10-14 days postdose)
  The HR will be measured by ECG.
Part 1: Change from Baseline in PR Interval | Baseline, 3, 24, 72 hours and at follow-up (10-14 days postdose)
  The PR Intervals will be measured by ECG.
Part 1: Change from Baseline in QRS Interval | Baseline, 3, 24, 72 hours and at follow-up (10-14 days postdose)
  The QRS Intervals will be measured by ECG.
Part 1: Percentage of Participants with T-Wave Morphology Changes from Baseline | Baseline up to 72 hours postdose
  Percentage of participants with T-wave morphology (Normal T-wave, Flat T-waves, Notched T-wave (positive), Biphasic, Normal T-wave (negative), Notched T-wave (negative) changes will be noted.
Part 1: Percentage of Participants with U-Wave Presence | Baseline up to 72 hours postdose
  Percentage of participants with U-wave presence will be noted.
Part 2: Change from Baseline in QTc Interval | Baseline, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, and 24 hours postdose
  The QT interval corrected for heart rate (QTc interval) using Fridericia method will be measured by ECG.
Part 2: Change from Baseline in HR | Baseline, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, and 24 hours postdose
  The HR will be measured by ECG.
Part 2: Change from Baseline PR Interval | Baseline, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, and 24 hours postdose
  The PR Intervals will be measured by ECG.
Part 2: Change from Baseline QRS Interval | Baseline, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, and 24 hours postdose
  The QRS Intervals will be measured by ECG.
Part 2: Placebo Corrected Change from Baseline in HR | Baseline, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, and 24 hours postdose
  Placebo-corrected change from baseline in HR will be determined. The mean change from baseline in HR in placebo treatment will be subtracted from the mean change from baseline in JNJ-53718678 treatment at the same time point to generate placebo-corrected change from baseline in HR, which will be presented.
Part 2: Placebo Corrected Change from Baseline PR Interval | Baseline, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, and 24 hours postdose
  Placebo-corrected change from baseline in PR interval will be determined. The mean change from baseline in PR interval in placebo treatment will be subtracted from the mean change from baseline in JNJ-53718678 treatment at the same time point to generate placebo-corrected change from baseline in PR interval, which will be presented.
Part 2: Placebo Corrected Change from Baseline QRS Interval | Baseline, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, and 24 hours postdose
  Placebo-corrected change from baseline in QRS interval will be determined. The mean change from baseline in QRS interval in placebo treatment will be subtracted from the mean change from baseline in JNJ-53718678 treatment at the same time point to generate placebo-corrected change from baseline in QRS interval, which will be presented.
Part 2: Number of Participants with Categorical Outliers for QTc Interval | Baseline up to 24 hours postdose
  Number of Participants with categorical outliers defined as QTc interval values greater than (>)450 and lesser than or equal to (<=) 480 milliseconds (ms), >480 and <=500 ms, and >500 ms at any time point and change from baseline QTc >30 ms and <=60 ms, and >60 ms will be determined.
Part 2: Number of Participants with Categorical Outliers for HR | Baseline up to 24 hours postdose
  Number of Participants with categorical outliers for HR will be determined for abnormality, where HR is abnormally low (<= 45 beats per minute [bpm]) and abnormally high (>= 120 bpm).
Part 2: Number of Participants with Categorical Outliers for PR Interval | Baseline up to 24 hours postdose
  Number of Participants with categorical outliers for PR interval will be determined for abnormality, where PR is abnormally high (>= 210 milliseconds [ms]).
Part 2: Number of Participants with Categorical Outliers for QRS Interval | Baseline up to 24 hours postdose
  Number of Participants with categorical outliers for QRS interval will be determined for abnormality, where QRS is abnormally low (<= 50 ms) and abnormally high (>=120 ms).
Part 2: Percentage of Participants with T-Wave Morphology Changes from Baseline | Baseline up to 24 hours postdose
  Percentage of participants with T-wave morphology (Normal T-wave, Flat T-waves, Notched T-wave (positive), Biphasic, Normal T-wave (negative), Notched T-wave (negative) changes will be noted.
Part 2: Percentage of Participants with U-Wave Presence | Baseline up to 24 hours postdose
  Percentage of participants with U-wave presence will be noted.
Part 1: Maximum Observed Plasma Concentration (Cmax) of JNJ-53718678 and its Metabolites (M5, M12, M19, and M37) | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours postdose
  Cmax is defined as the maximum observed plasma concentration. Cmax will be assessed for JNJ-53718678 and its metabolites (M5, M12, M19, and M37).
Part 1: Time to Reach Maximum Observed Plasma Concentration (Tmax) of JNJ-53718678 and its Metabolites (M5, M12, M19, and M37) | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours postdose
  Tmax is defined as actual sampling time to reach maximum observed plasma concentration. Tmax will be assessed for JNJ-53718678 and its metabolites (M5, M12, M19, and M37).
Part 1: Plasma concentration at 24 hours post dosing (C24h) of JNJ-53718678 and its Metabolites (M5, M12, M19, and M37) | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, and 24hours postdose
  C24h is defined as the plasma concentration at 24 hours post dosing. C24h will be assessed for JNJ-53718678 and its metabolites (M5, M12, M19, and M37).
Part 1: Area Under the Plasma Concentration-time Curve from Time 0 to 24 hours (AUC [0-24]) of JNJ-53718678 and its Metabolites (M5, M12, M19, and M37) | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, and 24 hours postdose
  AUC (0-24) is defined as the area under the plasma concentration-time curve from time 0 to 24 hours. AUC (0-24) will be assessed for JNJ-53718678 and its metabolites (M5, M12, M19, and M37).
Part 1: Area Under the Plasma Concentration-time Curve from Time Zero to the Time of Last Measurable Concentration (AUC [0-last]) of JNJ-53718678 and its Metabolites (M5, M12, M19, and M37) | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours postdose
  AUC(0-last) is defined as the area under the plasma concentration-time curve from time 0 to the time of the last measurable (non-below quantification level [non-BQL]) plasma concentration calculated by linear-linear trapezoidal summation. AUC [0-last] will be assessed for JNJ-53718678 and its metabolites (M5, M12, M19, and M37).
Part 1: Area Under the Plasma Concentration-time Curve from Time Zero to Infinity (AUC [0-infinity]) of JNJ-53718678 and its Metabolites (M5, M12, M19, and M37) | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours postdose
  AUC (0-infinity) is defined as the area under the plasma concentration vs. time curve from time 0 to infinite time, calculated as AUC (0-last) + Clast/ lambda (z), where Clast is the last observed measurable (non- BQL) plasma concentration. AUC (0-infinity) will be assessed for JNJ-53718678 and its metabolites (M5, M12, M19, and M37).
Part 1: Apparent Elimination Half-Life (T1/2) of JNJ- 53718678 and its Metabolites (M5, M12, M19, and M37) | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours postdose
  T1/2 is defined as apparent terminal elimination half-life and is calculated as 0.693/lambda(z) and will be assessed for JNJ-53718678 and its metabolites (M5, M12, M19, and M37).
Part 2: Maximum Observed Plasma Concentration (Cmax) of JNJ-53718678 and its Metabolites (M5, M12, M19, and M37) | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, and 24 hours postdose
  Cmax is defined as the maximum observed plasma concentration. Cmax will be assessed for JNJ-53718678 and its metabolites (M5, M12, M19, and M37).
Part 2: Time to Reach Maximum Observed Plasma Concentration (Tmax) of JNJ-53718678 and its Metabolites (M5, M12, M19, and M37) | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, and 24 hours postdose
  Tmax is defined as actual sampling time to reach maximum observed plasma concentration. Tmax will be assessed for JNJ-53718678 and its metabolites (M5, M12, M19, and M37).
Part 2: Area Under the Plasma Concentration-time Curve from Time 0 to 24 hours (AUC [0-24]) of JNJ-53718678 | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, and 24 hours postdose
  AUC (0-24) is defined as the area under the plasma concentration-time curve from time 0 to 24 hours. AUC (0-24) will be assessed for JNJ-53718678 and its metabolites (M5, M12, M19, and M37).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium